CLINICAL TRIAL: NCT03617627
Title: Self-management Intervention for Women With Chronic Pelvic Pain: a Randomized Controlled Trial
Brief Title: Self-management Program in Chronic Pelvic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Marie Carmen Valenza, PhD, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DF00800UG
Record Dates: First submitted 2018-07-31; First posted 2018-08-06 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Chronic Pelvic Pain
Keywords: chronic pain; women; self-management
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Patients will be included in a self-management intervention.
  Interventions: Behavioral: Self-management intervention
- Control group (No Intervention): Patients will receive a booklet with information.

INTERVENTIONS:
Behavioral: Self-management intervention — Self-management intervention will include presentation and discussion of various topics regarding chronic pain mechanisms and pain self-monitoring. The intervention will also incorporate a task-oriented approach focused on relevant activities in order to acquire coping skills.
  Arms: Experimental group

SUMMARY:
Chronic pelvic pain is a serious health condition with an estimated prevalence of 15% women worldwide.Treatment is a challenge given the different pain generators described. It is important to develop self-management interventions to reduce the frustration associated with its management.

DETAILED DESCRIPTION:
Chronic pelvic pain is defined as non-cyclic pain lasting for 6 or more months, that localizes to the anatomic pelvis, anterior abdominal wall at or below the umbilicus, the lumbosacral back, or the buttocks and is of sufficient severity to cause functional disability or lead to medical care. It can occur continuously or intermittently, with intensity severe enough to limit activities of daily living. It is frequent in women. The primary aim of this study isto evaluate the efficacy of a self-management intervention, as compared with an educational booklet in improving health-related quality of life and coping strategies, occupational performance, activity level and psycho-emotional symptoms in women with chronic pelvic pain.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic pelvic pain with at least 6 months of evolution

Exclusion Criteria:

* Active urogenital infection
* Pregnancy
* Cancer
* Dementia
* A surgical intervention involving lumbo-pelvic region over the past year

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2018-07-23 (Actual); Primary Completion 2018-10-21 (Actual); Study Completion 2019-04-29 (Actual)

PRIMARY OUTCOMES:
Perceived health-related quality of life | Change from baseline health-related quality of life at 7 weeks
  Health-related quality of life will be assessed using the EuroQol-5D. This scale consists of a descriptive system and the EQ visual analogue scale. The descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, oain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, extreme problems. Higher scores indicate more problems. In the visual analogue scale the patient rate the pain from 100 (best imaginable health state) to 0 (worst imaginable health state). Higher values represent a better health state.
Change in coping strategies | Change from baseline coping strategies at 7 weeks
  Coping strategies will be evaluated using the Coping Strategies Questionnaire (CSQ). It assesses eight different coping strategies for pain which describe two types of coping: adaptive coping (diverting Attention, coping self-statements, ignoring sensations, reinterpreting pain sensation, hoping and cognitive distracting) and maladaptive coping (catastrophizing, and faithing and praying). Participants score each item using a 7-point scale to indicate how often they use that strategy to manage their pain (0 never, 3 sometimes, and 6 always)

SECONDARY OUTCOMES:
Change in performance of activities | Change from baseline self-perceived performance at 7 weeks
  Canadian Occupational Performance Measure will be used to evaluate changes in patient's self-perception over time including performance and satisfaction scored from 0 to 10. Higher values represented improvement on perceived performance and satisfaction
Change in activity levels | Change from baseline self-reported activity levels at 7 weeks
  Activity levels will be evaluated with the International Physical Activity Questionnaire. It assess the frequency and time spent on vigorous, moderate-intensity activities and walking time for each category. Higher values indicate higher activity levels.
Change in anxiety levels. | Change from baseline anxious symptoms at 7 weeks
  Anxiety will be evaluated using the Beck Anxiety Inventory. It contains 21 questions, each answer being scored on a scale value of 0 (not at all) to 3 (severely). Higher total scores indicate more severe anxiety symptoms.
Change in depressive symptoms | Change from baseline depressive symptoms at 7 weeks
  Depression will be evaluated using the Beck Depression Inventory. It contains 21 questions, each answer being scored on a scale value of 0 (not at all) to 3 (severely). Higher total scores indicate severe depressive symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Marie Carmen Valenza, phD, Principal Investigator — Universidad de Granada
Locations (1):
- Department of Physical Therapy, Granada, Spain

IPD SHARING:
Plan to Share IPD: Undecided